CLINICAL TRIAL: NCT01338727
Title: Breastfeeding Education and Support Trial for Obese Women (BESTOW)
Acronym: BESTOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Rafael Pérez-Escamilla, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H06-009; DF05-015 (Other Grant/Funding Number: The Donaghue Foundation)
Record Dates: First submitted 2011-04-06; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Exclusive Breastfeeding; Breastfeeding Initiation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breastfeeding Peer Counseling (Experimental)
  Interventions: Behavioral: Breastfeeding Peer Counseling
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Breastfeeding Peer Counseling — 3 Prenatal visits, daily in-hospital visits, 11 postpartum home visits.
  Other Names: BESTOW
  Arms: Breastfeeding Peer Counseling

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a specialized exclusive breastfeeding education and support program targeting obese, pregnant, low-income women in Hartford, CT. Specifically, the investigators will evaluate the impact of the intervention on exclusive and partial breastfeeding rates at birth, 1, 3 and 6 months pp. Secondary aims of this study are: a) to characterize postpartum weight loss patterns and blood pressure values of obese women, by study group; and b) to evaluate potential differences in infant morbidity (diarrhea, otitis media and rehospitalization), by study group.

ELIGIBILITY:
Inclusion Criteria:

* obese (prepregnant BMI 27.0 or greater)
* pregnant women delivering at Hartford Hospital
* no more than 34 weeks gestation
* considering breastfeeding this child
* low income (<185% Federal poverty level)
* planning to remain in the greater Hartford area for 6 months postpartum
* must have access to a telephone for follow-up interviews
* delivery of a healthy, term, singleton

Exclusion Criteria:

* HIV positive or having other conditions which interfere with exclusive breastfeeding
* Infant admitted to the Neonatal Intensive Care Unit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Exclusive Breastfeeding Rate | 3 months postpartum

SECONDARY OUTCOMES:
Breastfeeding Rate | 3 months postpartum
Breastfeeding Initiation Rate | For the duration of the hospital stay, average equals 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Pérez-Escamilla, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Chapman DJ, Morel K, Bermudez-Millan A, Young S, Damio G, Perez-Escamilla R. Breastfeeding education and support trial for overweight and obese women: a randomized trial. Pediatrics. 2013 Jan;131(1):e162-70. doi: 10.1542/peds.2012-0688. Epub 2012 Dec 3. PMID 23209111